CLINICAL TRIAL: NCT04419194
Title: Association Between Climatic Factors and Hospital Admissions for Pulmonary Embolism: Time Series Study in China Between Years 2014 to 2019.
Brief Title: Effect of Climatic Factors on the Seasonal Fluctuation of Pulmonary Embolism
Status: Completed | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PUMCH-PE-Climatic factors
Record Dates: First submitted 2020-06-04; First posted 2020-06-05 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-05

CONDITIONS: Pulmonary Embolism
Keywords: Pulmonary Embolism; Climate
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observation: Observation

SUMMARY:
To estimate the risks of daily hospital admissions for pulmonary embolism associated with short term exposure to climatic factors (temperature, precipitation, air pressure, sunshine duration, relative humidity, wind speed, and ambient fine particulate matter [aerodynamic diameter ≤2.5 μm; PM2.5]) in China.

DETAILED DESCRIPTION:
Hospital admissions for pulmonary embolism were identified based on the primary diagnosis. The central adjudication committee at Peking Union Medical College Hospital (Beijing, China) reviewed all medical and death records and determined the final diagnosis. Two adjudication committee members verified events independently, and discrepancies were resolved by discussion involving additional committee members.For each admission, we extracted data on the date of admission, sex, age, and location of the patient from hospital information system.

All the data of daily meteorological variables for the same period, including temperature variables (°C) (the min, max and mean temperature), relative humidity (%), air pressure (hPa), precipitation (mm), wind speed (m/s) and sunshine duration (h), were collected from the China Meteorological Data Sharing Service System (http://www.escience.gov.cn/metdata/page/index.html). The data on PM2.5 levels in each city was collected from the National Air Pollution Monitoring System.

An overdispersed generalised additive model was used to estimate associations between climatic factors and pulmonary embolism admissions. A distributed lag non-linear model (DLNM) was employed to examine their lagged effects.

ELIGIBILITY:
Inclusion Criteria:

* Males and females.
* With a primary diagnosis of pulmonary embolism based on clinical symptoms, with or without radiologic features.

Exclusion Criteria:

* Lack of important data.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed as pulmonary embolism who meet the inclusion criteria above.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2014-07-31 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Incidence of pulmonary embolism | From July 31, 2014 to July 31, 2019
  Daily counts of hospital admissions for primary diagnoses of pulmonary embolism among different demographic groups were used to estimate the associations between climatic factors and morbidity.

CONTACTS AND LOCATIONS:
Overall Officials: Shi Juhong, M.D, Study Chair — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China